CLINICAL TRIAL: NCT02477384
Title: Randomised Trial of 8mm Transjugular Intrahepatic Portosystemic Shunt Versus Endoscopic Variceal Ligation Plus Propranolol for Prevention of Variceal Rebleeding
Brief Title: 8mm-TIPS Versus Endoscopic Variceal Ligation (EVL) Plus Propranolol for Prevention of Variceal Rebleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8mm-TIPS
Record Dates: First submitted 2015-06-15; First posted 2015-06-22 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8mm-TIPS (Active Comparator): Patients in this group would underwent TIPS placement with 8mm-diameter ePTFE-covered stents.
  Interventions: Procedure: 8mm-TIPS; Device: 8mm ePTFE-covered stent
- EVL plus propranolol (Active Comparator): Patients in this group would underwent sequential endoscopic variceal ligation and propranolol treatment.
  Interventions: Procedure: Endoscopic variceal ligation; Drug: Propranolol

INTERVENTIONS:
Procedure: 8mm-TIPS
  Arms: 8mm-TIPS
Procedure: Endoscopic variceal ligation
  Arms: EVL plus propranolol
Drug: Propranolol
  Arms: EVL plus propranolol
Device: 8mm ePTFE-covered stent
  Arms: 8mm-TIPS

SUMMARY:
The aim of this study was to conduct a prospective randomized trial to compare TIPS with 8mm expanded polytetrafluoroethylene(ePTFE)-covered stents and endoscopic variceal ligation plus propranolol for the prevention of recurrent esophageal variceal bleeding.

DETAILED DESCRIPTION:
For the prevention of recurrent esophageal variceal bleeding, previous clinical studies and meta-analysis show that patients treated with transjugular intrahepatic portosystemic shunt (TIPS) have lower rebleeding rates compared with endoscopic therapy. However, TIPS is associated with higher rates of portosystemic encephalopathy and does not show survival benefit. TIPS with a small-diameter may achieve sufficient portal decompression and reduce the incidence of hepatic encephalopathy. The aim of this study was to conduct a prospective randomized trial to compare TIPS with 8mm ePTFE-covered stents and endoscopic variceal ligation plus propranolol for the prevention of recurrent esophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis
2. Patients who had bled from esophageal varices (≥5days and ≤28days)
3. Child-Pugh B or Child-Pugh C≤13

Exclusion Criteria:

1. THE presence of gastric varices
2. Non-cirrhotic portal hypertension
3. Portal vein thrombosis
4. The history of hepatic encephalopathy
5. Total bilirubin ≥51.3 umol/L
6. Previous treatment of TIPS or surgery
7. Proven malignancy including hepatocellular carcinoma
8. Contraindications to TIPS、EVL or propranolol
9. End-stage renal disease under renal replacement therapy;
10. Cardiorespiratory failure
11. Pregnancy or patients not giving informed consent for endoscopic procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Variceal rebleeding rate | 3 years
  Analysis

SECONDARY OUTCOMES:
Hepatic encephalopathy rate | 3 years
  Analysis
Number of participants with improving or worsening hepatic function | 3 years
  Analysis
TIPS dysfunction rate | 3 years
  Analysis
The incidence of complications | 3 years
  Analysis
Number of participants with improving or worsening quality of life | 3 years
  Analysis
Mortality rate | 3 years
  Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Wang X, Liu G, Wu J, Xiao X, Yan Y, Guo Y, Yang J, Li X, He Y, Yang L, Luo X. Small-Diameter Transjugular Intrahepatic Portosystemic Shunt versus Endoscopic Variceal Ligation Plus Propranolol for Variceal Rebleeding in Advanced Cirrhosis. Radiology. 2023 Aug;308(2):e223201. doi: 10.1148/radiol.223201. PMID 37606572
- [Derived] Simonetti RG, Perricone G, Robbins HL, Battula NR, Weickert MO, Sutton R, Khan S. Portosystemic shunts versus endoscopic intervention with or without medical treatment for prevention of rebleeding in people with cirrhosis. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD000553. doi: 10.1002/14651858.CD000553.pub3. PMID 33089892